CLINICAL TRIAL: NCT06845436
Title: Effects of Combined High Intensity Interval Training and Resistance Training on Body Composition, Blood Pressure, and Cardiorespiratory Fitness in Obese Hypertensive Men
Brief Title: Effects of Combined High Intensity Interval Training and Resistance Training
Acronym: Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Ahmad Saied Mohammad, Dr, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCBR-430/2025
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
Keywords: hypertension.; obesity; High Intensity Interval Training; resistance training; blood pressure
MeSH Terms: conditions — Hypertension; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Combined exercise group subjects will undergo weekly three sessions of both HIIT and resistance training for sixteen weeks. The HIIT session will involve four four-minute high-intensity intervals with an intensity of at 80-95% of the HRmax interspersed with two-minute active recovery intervals with intensity of 40% to 60% of the HRmax. The resistance training session will be composed of eight exercises perform 3 sets of 8-12 repetitions with an intensity of 80% of the subject's estimated 1-RM. The HIIT only group perform 12 weeks of HIIT only.
  Interventions: Behavioral: Exercise
- control group (Other): The control group subjects will be instructed not to change their usual daily physical activities routine and instructed to abstain from practicing any exercise regimens during the 12-week study period.
  Interventions: Other: routine physical activity

INTERVENTIONS:
Behavioral: Exercise — Combined exercise group subjects will undergo weekly three sessions of both HIIT and resistance training for sixteen weeks. The HIIT session will involve four four-minute high-intensity intervals with an intensity of at 80-95% of the HRmax interspersed with two-minute active recovery intervals with intensity of 40% to 60% of the HRmax.
  Arms: study group
Other: routine physical activity — The control group subjects will be instructed not to change their usual daily physical activities routine and instructed to abstain from practicing any exercise regimens during the 12-week study period.
  Arms: control group

SUMMARY:
Background: Hypertension has long been considered as a major risk factor for cardiovascular disease representing a high public health concern.

Objectives: the purpose of this study is to evaluate the effects of combined HIIT and resistance training on body composition, blood pressure, and cardiorespiratory fitness in obese hypertensive men.

Methods: This study will make use of sixty obese hypertensive men aged 40 to 60 years. All participants meeting the eligibility criteria will be assigned to one of three groups; combined HIIT and resistance group, HIIT only group or control group. Combined exercise group subjects will undergo weekly three sessions of both HIIT and resistance training for sixteen weeks. The HIIT session will involve four four-minute high-intensity intervals with an intensity of at 80-95% of the HRmax interspersed with two-minute active recovery intervals with intensity of 40% to 60% of the HRmax. The resistance training session will be composed of eight exercises perform 3 sets of 8-12 repetitions with an intensity of 80% of the subject's estimated 1-RM. The HIIT only group perform 12 weeks of HIIT only. The control group subjects will be instructed not to change their usual daily physical activities routine and instructed to abstain from practicing any exercise regimens during the 12-week study period. Body composition measures, blood pressure and VO2peak will be assessed at baseline and at the end of the study period.

Results: All the outcome variables will be assessed at baseline and 12 weeks following the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* men aged between 40 and 60 years old,
* have been diagnosed with clinical stage 1 or 2 hypertension,
* being obese with body mass index more than 30 kg/m2
* physically inactive

Exclusion Criteria:

* musculoskeletal problems that may limit their ability to participate in resistance or HIIT programs
* diabetes mellitus
* a history of respiratory or chronic heart disease

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — male
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
blood pressure in mmhg | 12 weeks
peak oxygen consumption in ml/kg/min | 12 weeks
body weight in Kg | 12 weeks
body mass index in kg/m2 | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sattam bin Abdulaziz University, Riyadh, Alkharj, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No